CLINICAL TRIAL: NCT06085833
Title: ARTIDIS Nanomechanical Generated Measurements for Early Breast Lesions (ANGEL)
Brief Title: ARTIDIS Nanomechanical Generated Measurements for Early Breast Lesions
Acronym: ANGEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ARTIDIS AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ART-BrC-0102
Record Dates: First submitted 2023-04-28; First posted 2023-10-17 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Breast biopsy; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Masking Description: The sponsor is blinded toward the pathological diagnosis of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Human subjects requiring breast biopsy (Other): All patients referred to participating study sites for a core needle or vacuum-assisted breast biopsy are eligible for this study. Upon consent, a diagnostic biopsy will be measured by the sponsor's device before returning to the standard of care pathway.
  Interventions: Diagnostic Test: Nanomechanical Phenotype Test

INTERVENTIONS:
Diagnostic Test: Nanomechanical Phenotype Test — The ARTIDIS ART-1 device is an in-vitro diagnostic device based on Atomic Force Microscope (AFM) technology. The ART-1 device uses a probe to measure the nanomechanical phenotype of tissue components. ARTIDIS nanomechanical phenotype measurements are performed on fresh tissue after it is collected via biopsy or resection.

SUMMARY:
This prospective, blinded, single-arm study aims to test the performance of nanomechanical phenotype in predicting tumor type, tumor aggressiveness, and neoadjuvant treatment response compared to the gold standard of histopathological assessment. The study involves patients with suspicious breast lesions who will undergo a breast biopsy procedure indicated by standard of care. The nanomechanical phenotype will be measured on the freshly obtained breast biopsies or tissue from breast surgeries.

DETAILED DESCRIPTION:
Objective: To test the performance of nanomechanical phenotype tests in predicting tumor type, tumor aggressiveness, and neoadjuvant treatment response, compared to the gold standard of histopathological assessment on testing suspicious lesions.

Study Design:

This is a multi-center, blinded, single-arm study designed to collect nanomechanical signature measurement data of biopsy material taken for clinical diagnostic purposes in subjects referred for breast biopsy. Routine demographic, diagnostic and treatment data will be collected, as well as response evaluations. Subjects with a benign biopsy will be followed for a maximum of 30 days, while subjects diagnosed with breast cancer will be kept in active, routine, clinical follow-up with information collected twice yearly for the first two years and annually for years three to ten. Intermediate treatment biopsies or tissue samples from surgery may be collected at participating sites where they are performed routinely as standard of care (SOC).

All patients referred to participating study sites for a core needle or vacuum-assisted breast biopsy may be eligible for this study. All patients will be asked for written, informed consent for de-identified tissue and data collection on disease, histology characteristics, outcome, on disease related patent information, and patient reported outcomes.

The 2nd tissue core or representative core biopsies taken from the study subjects will be further investigated with the ARTIDIS platform and subsequently re-entered into the routine pathological analysis within the same day. Only two biopsies will be assessed per ART-1 device per day. One in the morning and one in the afternoon to ensure that the diagnostic biopsy can be reentered into the routine pathological analysis. The ARTIDIS measured biopsies will be marked to identify the orientation of the biopsy in the ART-1 device before re-entering the routine pathological analysis.

For malignant and benign lesions, follow up data will be extracted from the electronic medical record, as well as standard email/phone contacts performed by the study coordinator.

In order to assess the diagnostic performance of the proposed new method, it will be compared to the current gold standard. The participants cannot be randomized by study subjects with cancer vs. non cancer study subjects and will attempt to accrue a cohort representing a range of diagnostic outcomes in order to obtain a reasonable assessment of diagnostic performance.

Participants:

Patients with suspicious lesions who are referred for biopsy following routine mammography, ultrasound, MRI, and/or clinical evaluation.

Eligible subjects will be identified from each site's pool of patients by study investigators and the research team. Subjects will be asked to participate, interviewed and follow-up by explaining the possible benefit for future patients. Patients' advocates will participate in promotion of the study, as well as development of new strategies for recruitment if necessary.

Follow-up will be done by phone and/or email after consent according to study timelines, underlining future benefits of participation for other patients.

Outcome Measures:

The outcome measures will be the performance of nanomechanical phenotype tests in predicting tumor type, tumor aggressiveness, and neoadjuvant treatment response, compared to the gold standard of histopathological assessment.

Data Analysis:

Data will be analyzed using appropriate statistical methods to compare the performance of the nanomechanical phenotype test with the gold standard histopathological assessment. The full analysis set will consist of all patients, for whom both classifications of the core biopsy material are available, the one obtained from the ARTIDIS ART-1 device and the one from classical histopathological assessment.

Conclusion:

This study aims to determine the effectiveness of the nanomechanical phenotype test in predicting tumor type, tumor aggressiveness, and neoadjuvant treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Ability to understand and the willingness to sign a written informed consent.
* Indication for breast biopsy for diagnostic purposes
* ECOG performance status of 0 to 3.

Exclusion Criteria:

* Conditions that, in the investigator's opinion, might indicate that the subject is not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2706 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
ARTIDIS as a sensitive diagnostic tool | Read-out on day 30
  Variable, indicating a correct classification of patients' core biopsy material as malignant with the Nanomechanical Phenotype measurement in comparison to histopathological assessment as gold-standard.
ARTIDIS as a specific diagnostic tool | Read-out on day 30
  Variable, indicating a correct classification of patients' biopsy material as benign with the ARTIDIS Nanomechanical Phenotype measurement in comparison to histopathological assessment as gold-standard.

SECONDARY OUTCOMES:
ARTIDIS as an aid subtyping breast cancer | Read-out on day 30
  Diagnostic value (sensitivity) of subtype classification of invasive breast cancer with ARTIDIS Nanomechanical Phenotype Measurement compared to classical histopathology.
ARTIDIS imminent progression test as an indicator of local & regional progression | Read-out at 6 Months and annually up to 10 years
  Determine the ARTIDIS test's ability to detect local and regional progression at the time of diagnosis
ARTIDIS imminent progression test as an indicator of distant progression | Read-out at 6 Months and annually up to 10 years
  Determine the ARTIDIS test's ability to detect distant progression at the time of diagnosis
ARTIDIS imminent aggressiveness rating as a predictor of the pathological treatment response for patients receiving Neoadjuvant Treatment (NAT). | Read out at surgery
  Determine how well the ARTIDIS imminent aggressiveness rating predicts complete pathological treatment response at surgery for patients receiving Neoadjuvant Treatment.
ARTIDIS imminent aggressiveness rating as a predictor of the radiological treatment response for patients receiving Neoadjuvant Treatment (NAT). | Read out at surgery
  Determine how well the ARTIDIS imminent aggressiveness rating predicts radiological treatment response at the end of Neoadjuvant Treatment for patients receiving Neoadjuvant Treatment.
ARTIDIS ARTIDIS aggressiveness rating as a predictor of local recurrence-free survival time. | Read-out annually up to 10 years
  Determine the ability of the ARTIDIS aggressiveness rating to discriminate between patients with a high risk of recurrence and those with a low risk, adjusted for the applied cancer treatment.
ARTIDIS ARTIDIS aggressiveness rating as a predictor of disease-free survival time. | Read-out annually up to 10 years
  Determine the ability of the ARTIDIS aggressiveness rating to discriminate between patients with a high risk of suffering from further disease and those with a low risk, adjusted for the applied cancer treatment.
ARTIDIS ARTIDIS aggressiveness rating as a predictor of overall survival. | Read-out annually up to 10 years
  Determine the ability of the ARTIDIS aggressiveness rating to discriminate between patients with a high risk of dying from any cause and those with a low risk, adjusted for the applied cancer treatment.
ARTIDIS potential in distinguishing benign from malignant lesions with nanomechanical profiles in relation to different tissue sources. | Read-out on day 30
  Variable, indicating a correct classification of patients' biopsy material by ARTIDIS Nanomechanical Phenotype Measurement in comparison to Histopathology in relation to different tissue sources (e.g. CNB, VAB, MRI guided biopsy etc.).

OTHER OUTCOMES:
Exploratory Objective 1: ARTIDIS as an aid for diagnostic efficacy for radiologically assessed breast lesions. | Read-out on day 30
  Diagnostic value (sensitivity) of BI-RADS 4 assessment in combination with Nanomechanical Phenotype Measurement or without Nanomechanical Phenotype Measurement with histopathological assessment as gold-standard.
Exploratory Objective 2: ARTIDIS as an aid for radiologist to improve the reliability of BI-RADS classification. | Read-out on day 30
  Diagnostic value (sensitivity) of all BI-RADS assessments in combination with Nanomechanical Phenotype Measurement or without Nanomechanical Phenotype Measurement with histopathological assessment as gold-standard.
Exploratory Objective 3: ARTIDIS potential in improving time to treatment initiation for patients with a malignant breast lesion in comparison to standard workflow. | Read-out during the follow-up visits on month 6, month 12, and then annually up to 10 years
  Measurement of reduction of time to treatment initiation for patients with a high aggressive malignant lesion without ARTIDIS imminent aggressiveness measurement compared to time to treatment initiation with ARTIDIS imminent aggressiveness measurement via health care navigator interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Thompson, MD, Principal Investigator — Baylor College of Medicine
Locations (5):
- United States (3):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Clinic - Mays Clinic, Houston, Texas
- Hospital Universitario Vall d'Hebron, Barcelona, Barcelona, Spain
- Claraspital, Basel, Basel, Switzerland

REFERENCES:
- [Background] Plodinec M, Loparic M, Monnier CA, Obermann EC, Zanetti-Dallenbach R, Oertle P, Hyotyla JT, Aebi U, Bentires-Alj M, Lim RY, Schoenenberger CA. The nanomechanical signature of breast cancer. Nat Nanotechnol. 2012 Nov;7(11):757-65. doi: 10.1038/nnano.2012.167. Epub 2012 Oct 21. PMID 23085644